CLINICAL TRIAL: NCT05533034
Title: Personalized Home Respiratory Rehabilitation Program for Subjects With Systemic Sclerosis With Early Lung Disease: Pilot Feasibility Study
Brief Title: Personalized Home Respiratory Rehabilitation Program for Subjects With Systemic Sclerosis With Early Lung Disease
Acronym: SCLERESPIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210260; 2020-A03551-38 (Other: France : ANSM)
Record Dates: First submitted 2022-07-07; First posted 2022-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis; Lung disease; Rehabilitation; Respiratory deficiencies; Feasibility study
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home based exercises (Experimental): 1 supervised session in the outpatient rehabilitation department with respiratory, aerobic and muscles strengthening exercises, followed by 3 months of self-manage personalized home exercises program. Cardiac frequency and adherence to exercise will be monitored using an activity tracker (Garmin© watch).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — * 1 supervised session of rehabilitation, including a cardiac stress test (to define maximal intensity for aerobic activities), aerobic activity with interval training of moderate and progressive intensity (walking), and respiratory exercise using a volumetric spirometer, and strengthening exercises for lower and upper limbs.
  * 3 months of self-managed home exercises. Patients will be asked to use a tracker activity when performing home exercises to self-monitor cardiac frequency and to assess their adherence.
  Other Names: Personalized home exercises program

SUMMARY:
Systematic sclerosis (SSc) is a potentially severe disease characterized by various visceral involvements including lung. The investigators hypothesize that a respiratory rehabilitation program specifically designed for people with systematic sclerosis with early lung disease could help to decrease respiratory deficiencies, improve aerobic capacity and prevent activity limitations and participation restrictions.

Before testing the effectiveness of such a program, a pilot study is needed to assess its feasibility and optimize its content.

Participants will have 1 supervised session in the outpatient rehabilitation department. Each patient will then perform the home personalized exercises program for 3 months.

The feasibility of the program will be assessed at 3 months using patients' adherence to the program (assessed by the number of lost to follow-up, the number of questionnaires not completed, the amount of aerobic activity and the amount of home personalized exercises, treatment burden, adverse effects and quality of life.

DETAILED DESCRIPTION:
SSc is responsible for a reduced life expectancy. The prognosis depends on the presence of severe visceral damage and more particularly on the presence of interstitial lung damage, pulmonary arterial hypertension or specific cardiac damage which represent the 3 main causes of mortality in SSc.

The importance of rehabilitation in SSc has been confirmed by the latest INSERM Collective Expertise 2019). The objectives of functional rehabilitation in SSc are to prevent and/or reduce the specific (cutaneous, oral, cardiorespiratory, musculoskeletal) and non-specific (exercise deconditioning, fatigue, anxiety and depression) impairments frequently characterizing the evolution of the disease. Based on the latest practice recommendations for the diagnosis and treatment of idiopathic pulmonary fibrosis, people with a confirmed diagnosis of idiopathic pulmonary fibrosis and significant exercise and activity limitations should follow a respiratory rehabilitation program.

The value of a specific respiratory rehabilitation program for people with SSc is then a matter of interest. A pilot study is needed to assess the feasibility and optimize the content of a rehabilitation program. The investigators aimed to study the feasibility of a personalized home-based respiratory rehabilitation program in people with SSc with early lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis according to ACR/EULAR 2013 criteria
* Lung involvement, with FCV > 70% on PFT

Exclusion Criteria:

* Inability to understand French
* Pregnancy or breastfeeding
* Arterial pulmonary hypertension > 35 mmHg and unexplained dyspnoea or arterial pulmonary hypertension > 40 mmHg
* Major musculoskeletal impairment incompatible with physical activity
* other pulmonary disease decreasing FCV
* Pathological EKG
* Oxygen saturation at rest or during physical activity < 90%
* FCV < 70%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of lost to follow up patients | 3 months
  Adherence to treatment
Number of uncompleted questionnaires | 3 months
  Adherence to treatment
Amount of aerobic work recorded using a connected watch | 3 months
  Adherence to treatment / Amount of aerobic work recorded using a connected watch with heart rate monitor
Amount of exercises self-reported in a logbook | 3 months
  Adherence to treatment
Exercise Adherence Rating Scale (EARS) questionnaire | 3 months
  Adherence to treatment / Amount of exercises
Self-reported adherence | 3 months
  Adherence to treatment
Exercise Adherence Rating Scale (EARS) questionnaire | 3 months
  Adherence to treatment
Treatment burden assess by the Exercise Therapy Burden Questionnaire (ETBQ) | 3 months
  Adherence to treatment / Burden of program
Check-list to report side effects | 3 months
  Adherence to treatment

SECONDARY OUTCOMES:
Lung volume | Day of inclusion
  Pulmonary Function Testing (PFT) - Respiratory function / Variation between base line and 3 months
Lung volume | 3 months
  Pulmonary Function Testing (PFT) - Respiratory function / Variation between base line and 3 months
Diffusing capacity | Day of inclusion
  Pulmonary Function Testing (PFT) - Respiratory function / Variation between base line and 3 months
Diffusing capacity | 3 months
  Pulmonary Function Testing (PFT) - Respiratory function / Variation between base line and 3 months
Maximal oxygen consumption during a 6 minute walking test | Day of inclusion
  Aerobic capacity / Variation between base line and 3 months
Maximal oxygen consumption during a 6 minute walking test | 3 months
  Aerobic capacity / Variation between base line and 3 months
Saint Georges hospital questionnaire | Day of inclusion
  Activity limitations specific to respiratory function / Variation between base line and 3 months
Saint Georges hospital questionnaire | 3 months
  Activity limitations specific to respiratory function / Variation between base line and 3 months
Health Assessment Questionnaire (HAQ) | Day of inclusion
  Overall activity limitations / Variation between base line and 3 months
Health Assessment Questionnaire (HAQ) | 3 months
  Overall activity limitations / Variation between base line and 3 months
12-Items short form survey questionnaire (SF-12) | Day of inclusion
  Quality of life / Variation between base line and 3 months
12-Items short form survey questionnaire (SF-12) | 3 months
  Quality of life / Variation between base line and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Camille DASTE, MD, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP); Christelle NGUYEN, MD, PhD, Study Director — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Service de rééducation fonctionnelle, réadaptation de l'appareil locomoteur et Pathologies du Rachis - Cochin Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided